CLINICAL TRIAL: NCT04371419
Title: COVID-19 Health Messaging to Underserved Communities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Bureau of Economic Research, Inc. (Other)
Collaborators: Massachusetts General Hospital (Other); Stanford University (Other); Yale University (Other); Massachusetts Institute of Technology (Other); Harvard University (Other)
Responsible Party: Principal Investigator, Esther Duflo, Abdul Latif Jameel Professor of Poverty Alleviation and Development Economics, MIT; Co-Director, Abdul Latif Jameel Poverty Action Lab, National Bureau of Economic Research, Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2003000118
Record Dates: First submitted 2020-04-28; First posted 2020-05-01 (Actual); Results first posted 2021-07-27 (Actual); Last update posted 2021-07-27 (Actual); Status verified 2021-07

CONDITIONS: Coronavirus
MeSH Terms: conditions — Coronavirus Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (17):
- Control - CDC - Mask (Control) - Concordant (Experimental): Control Intro, CDC Social Distancing, Mask Control version delivered by minority doctor of same background as the recipient - other definitions are similar
  Interventions: Behavioral: Messaging
- Control - CDC - Mask (Control) - Discordant (Experimental): Control Intro, CDC Social Distancing, Mask Control version delivered by majority doctor of different background as the recipient - other definitions are similar
  Interventions: Behavioral: Messaging
- Control - MGH - Mask (Control) - Concordant (Experimental): Control Intro, MGH Social Distancing, Mask Control version delivered by concordant doctor
  Interventions: Behavioral: Messaging
- Control - MGH - Mask (Control) - Discordant (Experimental): Control Intro, MGH Social Distancing, Mask Control version delivered by discordant doctor
  Interventions: Behavioral: Messaging
- Ack. Discrimination- MGH - Mask (Control) - Concordant (Experimental): Introduction Acknowledges past discrimination, MGH doctor talks about Social Distancing, Mask Control all by concordant MD
  Interventions: Behavioral: Messaging
- Ack. Discrimination- MGH - Mask (Control) - Discordant (Experimental): Introduction Acknowledges past discrimination, MGH doctor talks about Social Distancing, Mask Control all by discordant MD
  Interventions: Behavioral: Messaging
- Ack. econ. circumstance- MGH - Mask (Control ) Concordant (Experimental): Intro econ. circumstance -MGH - Mask (Control ) Concordant
  Interventions: Behavioral: Messaging
- Ack. econ. circumstance - MGH - Mask (Control ) Discordant (Experimental)
  Interventions: Behavioral: Messaging
- Control Intro - CDC - Mask (antiStigma) Concordant (Experimental): Control Intro - CDC - Mask (antiStigma) Concordant messenger
  Interventions: Behavioral: Messaging
- Control Intro - CDC - Mask (antiStigma) Discordant (Experimental): Control Intro - CDC - Mask (antiStigma) discordant messenger
  Interventions: Behavioral: Messaging
- Control - MGH - MaskS (antiStigma) Concordant messenger (Experimental): Control - MGH - MaskS (antiStigma) Concordant sender
  Interventions: Behavioral: Messaging
- Control- MGH-MaskS (antiStigma) Discordant messenger (Experimental): Control - MGH - MaskS (antiStigma) Discordant sender
  Interventions: Behavioral: Messaging
- Ack. Discrimination - MGH - MaskS (antiStigma) Concordant (Experimental): Acknowledge Discrimination - MGH - MaskS (antiStigma) Concordant sender
  Interventions: Behavioral: Messaging
- Ack. Discrimination - MGH - MaskS (antiStigma) Discordant (Experimental): Acknowledge Discrimination - MGH - MaskS (antiStigma) Discordant sender
  Interventions: Behavioral: Messaging
- Ack. Econ Hardship- MGH - Mask (antiStigma) Concordant (Experimental): Acknowledge Econ Hardship- MGH - Mask (antiStigma) Concordant sender
  Interventions: Behavioral: Messaging
- Ack. Econ Hardship- MGH - Mask (antiStigma) Discordant (Experimental): Acknowledge Econ Hardship- MGH - Mask (antiStigma) discordant sender
  Interventions: Behavioral: Messaging
- Info later - Pure Control (Placebo Comparator): This group will not receive the videos but will receive information later.
  Interventions: Behavioral: Messaging

INTERVENTIONS:
Behavioral: Messaging — o The video messages each participant in one of the treatment groups sees will be randomized on the following dimensions. The different versions are clearly demarcated in the US Doctors Scripts document.
  * Racial or ethnic identity of the doctor delivering the messages: concordant vs. discordant identity to the subject.
  * Whether the message includes an acknowledgment of "elephant in the room" issues for each target group: trust in the medical system or fear of deportation.
  * Whether the social distancing component of the message is delivered by Dr. Birx of the CDC or recorded by the MGH physicians.
  * Whether individuals are given information about how representative individuals perceive mask wearers of color. This information comes from results of our nationally representative pilot survey.
  * Some individuals in a control group will see messages later.

SUMMARY:
Recent data have shown that covid19 is disproportionately infecting and killing African Americans and Latinx people in the United States. The aim of the study is to determine which messages are most effective at increasing knowledge and changing behaviors that can protect individuals and their communities from the virus. To accomplish this aim, we plan to recruit approximately 20,000 Hispanic and African-American individuals and randomly assign them to videos that vary either the sender or the framing of the message, while providing the relevant public health information.

DETAILED DESCRIPTION:
The following procedures will be followed. The research subjects will participate online.

1. Doctors from MGH who express interest in participating will record messages according to our scripts (US Doctors Script African American, US Doctors Script Latinx). They will be instructed to film several different versions each.
2. We will recruit a sample of Latinx and African American study participants from across the country through Lucid, an online survey firm that has access to a large subject pool.
3. Participants will first read a consent script and give us their informed consent (US Doctors Messaging Consent)
4. Participants will then navigate through the following steps

   1. Brief demographics survey questions (US Doctors Messaging Survey)
   2. Videos 1 and 2: Introduction, Acknowledgement, Social Distancing (US Doctors Script African American, US Doctors Script Latinx). Individuals in the control group will not see videos.
   3. Beliefs survey questions (US Doctors Messaging Survey)
   4. Video 3: Masks (US Doctors Script African American, US Doctors Script Latinx). Again, individuals in the control group will not see a video here.
   5. Main outcomes survey (US Doctors Messaging Survey)
   6. Control group is shown a version of all 3 videos at end (US Doctors Script African American, US Doctors Script Latinx).
5. The video messages each participant in one of the treatment groups sees will be randomized on the following dimensions. The different versions are clearly demarcated in the US Doctors Scripts document.

   1. Racial or ethnic identity of the doctor delivering the messages: concordant vs. discordant identity to the subject.
   2. Whether the message includes an acknowledgment of "elephant in the room" issues for each target group: trust in the medical system or fear of deportation.
   3. Whether the social distancing component of the message is delivered by Dr. Birx of the CDC or recorded by the MGH physicians.
   4. Whether individuals are given information about how representative individuals perceive mask wearers of color. This information comes from results of our nationally representative pilot survey.
   5. Some individuals in a control group will only see messages after all surveying has been completed.

ELIGIBILITY:
Inclusion Criteria: Hispanic and African-American adult individuals, men and women - oversample of those with less completed education Exclusion Criteria: children, those who do not identify as above

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14267 (Actual)
Dates: Start 2020-05-13 (Actual); Primary Completion 2020-05-24 (Actual); Study Completion 2020-05-26 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- JPAL North America, Cambridge, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Generally, economists will post code and de-identified data when the findings are published
Supporting Information: SAP, Analytic Code
Time Frame: Generally, social scientists post code and de-identified data when the findings are published
Access Criteria: To be determined, if published alongside the paper data and code may be gated.

REFERENCES:
- [Derived] Alsan M, Stanford FC, Banerjee A, Breza E, Chandrasekhar AG, Eichmeyer S, Goldsmith-Pinkham P, Ogbu-Nwobodo L, Olken BA, Torres C, Sankar A, Vautrey PL, Duflo E. Comparison of Knowledge and Information-Seeking Behavior After General COVID-19 Public Health Messages and Messages Tailored for Black and Latinx Communities : A Randomized Controlled Trial. Ann Intern Med. 2021 Apr;174(4):484-492. doi: 10.7326/M20-6141. Epub 2020 Dec 21. PMID 33347320

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Individuals were recruited throughout the United States by the survey company Lucid from 13 May to 26 May 2020. Only persons aged 18 years or older and self-identifying as Black or Latinx were eligible.
Pre-assignment Details: The trial sample was enrolled from 13 May 2020 through 26 May 2020. Of 35,987 persons screened, 20,925 were eligible for participation (15,062 who would have been eligible were excluded because the demographic quotas were met); 5,450 individuals did not consent or failed both basic attention checks, and 1,208 left the survey before randomization. Out of 14,267 participants enrolled and randomized,123 participants did not answer one or more baseline questions and were excluded from analysis.
Groups:
- Control - CDC - Mask (Control) - Concordant: Control Intro, CDC Social Distancing, Mask Control version delivered by minority doctor of same background as the recipient - other definitions are similar
  Messaging: o The video messages each participant in one of the treatment groups sees will be randomized on the following dimensions. The different versions are clearly demarcated in the US Doctors Scripts document.
  * Racial or ethnic identity of the doctor delivering the messages: concordant vs. discordant identity to the subject.
  * Whether the message includes an acknowledgment of "elephant in the room" issues for each target group: trust in the medical system or fear of deportation.
  * Whether the social distancing component of the message is delivered by Dr. Birx of the CDC or recorded by the MGH physicians.
  * Whether individuals are given information about how representative individuals perceive mask wearers of color. This information comes from results of our nationally representative pilot survey.
  * Some individuals in a control group will see messages later.
- Control - CDC - Mask (Control) - Discordant: Control Intro, CDC Social Distancing, Mask Control version delivered by majority doctor of different background as the recipient - other definitions are similar
  Messaging: o The video messages each participant in one of the treatment groups sees will be randomized on the following dimensions. The different versions are clearly demarcated in the US Doctors Scripts document.
  * Racial or ethnic identity of the doctor delivering the messages: concordant vs. discordant identity to the subject.
  * Whether the message includes an acknowledgment of "elephant in the room" issues for each target group: trust in the medical system or fear of deportation.
  * Whether the social distancing component of the message is delivered by Dr. Birx of the CDC or recorded by the MGH physicians.
  * Whether individuals are given information about how representative individuals perceive mask wearers of color. This information comes from results of our nationally representative pilot survey.
  * Some individuals in a control group will see messages later.
- Control - MGH - Mask (Control) - Concordant: Control Intro, MGH Social Distancing, Mask Control version delivered by concordant doctor
  Messaging: o The video messages each participant in one of the treatment groups sees will be randomized on the following dimensions. The different versions are clearly demarcated in the US Doctors Scripts document.
  * Racial or ethnic identity of the doctor delivering the messages: concordant vs. discordant identity to the subject.
  * Whether the message includes an acknowledgment of "elephant in the room" issues for each target group: trust in the medical system or fear of deportation.
  * Whether the social distancing component of the message is delivered by Dr. Birx of the CDC or recorded by the MGH physicians.
  * Whether individuals are given information about how representative individuals perceive mask wearers of color. This information comes from results of our nationally representative pilot survey.
  * Some individuals in a control group will see messages later.
- Control - MGH - Mask (Control) - Discordant: Control Intro, MGH Social Distancing, Mask Control version delivered by discordant doctor
  Messaging: o The video messages each participant in one of the treatment groups sees will be randomized on the following dimensions. The different versions are clearly demarcated in the US Doctors Scripts document.
  * Racial or ethnic identity of the doctor delivering the messages: concordant vs. discordant identity to the subject.
  * Whether the message includes an acknowledgment of "elephant in the room" issues for each target group: trust in the medical system or fear of deportation.
  * Whether the social distancing component of the message is delivered by Dr. Birx of the CDC or recorded by the MGH physicians.
  * Whether individuals are given information about how representative individuals perceive mask wearers of color. This information comes from results of our nationally representative pilot survey.
  * Some individuals in a control group will see messages later.
- Ack. Discrimination- MGH - Mask (Control) - Concordant: Introduction Acknowledges past discrimination, MGH doctor talks about Social Distancing, Mask Control all by concordant MD
  Messaging: o The video messages each participant in one of the treatment groups sees will be randomized on the following dimensions. The different versions are clearly demarcated in the US Doctors Scripts document.
  * Racial or ethnic identity of the doctor delivering the messages: concordant vs. discordant identity to the subject.
  * Whether the message includes an acknowledgment of "elephant in the room" issues for each target group: trust in the medical system or fear of deportation.
  * Whether the social distancing component of the message is delivered by Dr. Birx of the CDC or recorded by the MGH physicians.
  * Whether individuals are given information about how representative individuals perceive mask wearers of color. This information comes from results of our nationally representative pilot survey.
  * Some individuals in a control group will see messages later.
- Ack. Discrimination- MGH - Mask (Control) - Discordant: Introduction Acknowledges past discrimination, MGH doctor talks about Social Distancing, Mask Control all by discordant MD
  Messaging: o The video messages each participant in one of the treatment groups sees will be randomized on the following dimensions. The different versions are clearly demarcated in the US Doctors Scripts document.
  * Racial or ethnic identity of the doctor delivering the messages: concordant vs. discordant identity to the subject.
  * Whether the message includes an acknowledgment of "elephant in the room" issues for each target group: trust in the medical system or fear of deportation.
  * Whether the social distancing component of the message is delivered by Dr. Birx of the CDC or recorded by the MGH physicians.
  * Whether individuals are given information about how representative individuals perceive mask wearers of color. This information comes from results of our nationally representative pilot survey.
  * Some individuals in a control group will see messages later.
- Ack. Econ. Circumstance- MGH - Mask (Control ) Concordant: Intro econ. circumstance -MGH - Mask (Control ) Concordant
  Messaging: o The video messages each participant in one of the treatment groups sees will be randomized on the following dimensions. The different versions are clearly demarcated in the US Doctors Scripts document.
  * Racial or ethnic identity of the doctor delivering the messages: concordant vs. discordant identity to the subject.
  * Whether the message includes an acknowledgment of "elephant in the room" issues for each target group: trust in the medical system or fear of deportation.
  * Whether the social distancing component of the message is delivered by Dr. Birx of the CDC or recorded by the MGH physicians.
  * Whether individuals are given information about how representative individuals perceive mask wearers of color. This information comes from results of our nationally representative pilot survey.
  * Some individuals in a control group will see messages later.
- Control Intro - CDC - Mask (antiStigma) Concordant: Control Intro - CDC - Mask (antiStigma) Concordant messenger
  Messaging: o The video messages each participant in one of the treatment groups sees will be randomized on the following dimensions. The different versions are clearly demarcated in the US Doctors Scripts document.
  * Racial or ethnic identity of the doctor delivering the messages: concordant vs. discordant identity to the subject.
  * Whether the message includes an acknowledgment of "elephant in the room" issues for each target group: trust in the medical system or fear of deportation.
  * Whether the social distancing component of the message is delivered by Dr. Birx of the CDC or recorded by the MGH physicians.
  * Whether individuals are given information about how representative individuals perceive mask wearers of color. This information comes from results of our nationally representative pilot survey.
  * Some individuals in a control group will see messages later.
- Control Intro - CDC - Mask (antiStigma) Discordant: Control Intro - CDC - Mask (antiStigma) discordant messenger
  Messaging: o The video messages each participant in one of the treatment groups sees will be randomized on the following dimensions. The different versions are clearly demarcated in the US Doctors Scripts document.
  * Racial or ethnic identity of the doctor delivering the messages: concordant vs. discordant identity to the subject.
  * Whether the message includes an acknowledgment of "elephant in the room" issues for each target group: trust in the medical system or fear of deportation.
  * Whether the social distancing component of the message is delivered by Dr. Birx of the CDC or recorded by the MGH physicians.
  * Whether individuals are given information about how representative individuals perceive mask wearers of color. This information comes from results of our nationally representative pilot survey.
  * Some individuals in a control group will see messages later.
- Control - MGH - MaskS (antiStigma) Concordant Messenger: Control - MGH - MaskS (antiStigma) Concordant sender
  Messaging: o The video messages each participant in one of the treatment groups sees will be randomized on the following dimensions. The different versions are clearly demarcated in the US Doctors Scripts document.
  * Racial or ethnic identity of the doctor delivering the messages: concordant vs. discordant identity to the subject.
  * Whether the message includes an acknowledgment of "elephant in the room" issues for each target group: trust in the medical system or fear of deportation.
  * Whether the social distancing component of the message is delivered by Dr. Birx of the CDC or recorded by the MGH physicians.
  * Whether individuals are given information about how representative individuals perceive mask wearers of color. This information comes from results of our nationally representative pilot survey.
  * Some individuals in a control group will see messages later.
- Control- MGH-MaskS (antiStigma) Discordant Messenger: Control - MGH - MaskS (antiStigma) Discordant sender
  Messaging: o The video messages each participant in one of the treatment groups sees will be randomized on the following dimensions. The different versions are clearly demarcated in the US Doctors Scripts document.
  * Racial or ethnic identity of the doctor delivering the messages: concordant vs. discordant identity to the subject.
  * Whether the message includes an acknowledgment of "elephant in the room" issues for each target group: trust in the medical system or fear of deportation.
  * Whether the social distancing component of the message is delivered by Dr. Birx of the CDC or recorded by the MGH physicians.
  * Whether individuals are given information about how representative individuals perceive mask wearers of color. This information comes from results of our nationally representative pilot survey.
  * Some individuals in a control group will see messages later.
- Ack. Discrimination - MGH - MaskS (antiStigma) Concordant: Acknowledge Discrimination - MGH - MaskS (antiStigma) Concordant sender
  Messaging: o The video messages each participant in one of the treatment groups sees will be randomized on the following dimensions. The different versions are clearly demarcated in the US Doctors Scripts document.
  * Racial or ethnic identity of the doctor delivering the messages: concordant vs. discordant identity to the subject.
  * Whether the message includes an acknowledgment of "elephant in the room" issues for each target group: trust in the medical system or fear of deportation.
  * Whether the social distancing component of the message is delivered by Dr. Birx of the CDC or recorded by the MGH physicians.
  * Whether individuals are given information about how representative individuals perceive mask wearers of color. This information comes from results of our nationally representative pilot survey.
  * Some individuals in a control group will see messages later.
- Ack. Discrimination - MGH - MaskS (antiStigma) Discordant: Acknowledge Discrimination - MGH - MaskS (antiStigma) Discordant sender
  Messaging: o The video messages each participant in one of the treatment groups sees will be randomized on the following dimensions. The different versions are clearly demarcated in the US Doctors Scripts document.
  * Racial or ethnic identity of the doctor delivering the messages: concordant vs. discordant identity to the subject.
  * Whether the message includes an acknowledgment of "elephant in the room" issues for each target group: trust in the medical system or fear of deportation.
  * Whether the social distancing component of the message is delivered by Dr. Birx of the CDC or recorded by the MGH physicians.
  * Whether individuals are given information about how representative individuals perceive mask wearers of color. This information comes from results of our nationally representative pilot survey.
  * Some individuals in a control group will see messages later.
- Ack. Econ Hardship- MGH - Mask (antiStigma) Concordant: Acknowledge Econ Hardship- MGH - Mask (antiStigma) Concordant sender
  Messaging: o The video messages each participant in one of the treatment groups sees will be randomized on the following dimensions. The different versions are clearly demarcated in the US Doctors Scripts document.
  * Racial or ethnic identity of the doctor delivering the messages: concordant vs. discordant identity to the subject.
  * Whether the message includes an acknowledgment of "elephant in the room" issues for each target group: trust in the medical system or fear of deportation.
  * Whether the social distancing component of the message is delivered by Dr. Birx of the CDC or recorded by the MGH physicians.
  * Whether individuals are given information about how representative individuals perceive mask wearers of color. This information comes from results of our nationally representative pilot survey.
  * Some individuals in a control group will see messages later.
- Ack. Econ Hardship- MGH - Mask (antiStigma) Discordant: Acknowledge Econ Hardship- MGH - Mask (antiStigma) discordant sender
  Messaging: o The video messages each participant in one of the treatment groups sees will be randomized on the following dimensions. The different versions are clearly demarcated in the US Doctors Scripts document.
  * Racial or ethnic identity of the doctor delivering the messages: concordant vs. discordant identity to the subject.
  * Whether the message includes an acknowledgment of "elephant in the room" issues for each target group: trust in the medical system or fear of deportation.
  * Whether the social distancing component of the message is delivered by Dr. Birx of the CDC or recorded by the MGH physicians.
  * Whether individuals are given information about how representative individuals perceive mask wearers of color. This information comes from results of our nationally representative pilot survey.
  * Some individuals in a control group will see messages later.
- Info Later - Pure Control: This group will not receive the videos but will receive information later.
  Messaging: o The video messages each participant in one of the treatment groups sees will be randomized on the following dimensions. The different versions are clearly demarcated in the US Doctors Scripts document.
  * Racial or ethnic identity of the doctor delivering the messages: concordant vs. discordant identity to the subject.
  * Whether the message includes an acknowledgment of "elephant in the room" issues for each target group: trust in the medical system or fear of deportation.
  * Whether the social distancing component of the message is delivered by Dr. Birx of the CDC or recorded by the MGH physicians.
  * Whether individuals are given information about how representative individuals perceive mask wearers of color. This information comes from results of our nationally representative pilot survey.
  * Some individuals in a control group will see messages later.
Period: Overall Study
Arm/Group | Control - CDC - Mask (Control) - Concordant | Control - CDC - Mask (Control) - Discordant | Control - MGH - Mask (Control) - Concordant | Control - MGH - Mask (Control) - Discordant | Ack. Discrimination- MGH - Mask (Control) - Concordant | Ack. Discrimination- MGH - Mask (Control) - Discordant | Ack. Econ. Circumstance- MGH - Mask (Control ) Concordant | Ack. Econ. Circumstance - MGH - Mask (Control ) Discordant | Control Intro - CDC - Mask (antiStigma) Concordant | Control Intro - CDC - Mask (antiStigma) Discordant | Control - MGH - MaskS (antiStigma) Concordant Messenger | Control- MGH-MaskS (antiStigma) Discordant Messenger | Ack. Discrimination - MGH - MaskS (antiStigma) Concordant | Ack. Discrimination - MGH - MaskS (antiStigma) Discordant | Ack. Econ Hardship- MGH - Mask (antiStigma) Concordant | Ack. Econ Hardship- MGH - Mask (antiStigma) Discordant | Info Later - Pure Control
Started | 784 | 791 | 780 | 778 | 777 | 788 | 783 | 788 | 779 | 780 | 782 | 790 | 779 | 786 | 781 | 781 | 1617
Completed the Knowledge Questions (Participants who completed the knowledge questions and were included in the knowledge outcome analysis questions) | 663 | 669 | 673 | 664 | 666 | 683 | 664 | 679 | 670 | 655 | 656 | 692 | 664 | 687 | 652 | 652 | 1526
Completed (Participants completed the survey and were included in all analyses.) | 641 | 636 | 639 | 631 | 644 | 654 | 639 | 658 | 649 | 621 | 626 | 662 | 633 | 660 | 626 | 625 | 1450
Not Completed | 143 | 155 | 141 | 147 | 133 | 134 | 144 | 130 | 130 | 159 | 156 | 128 | 146 | 126 | 155 | 156 | 167

BASELINE CHARACTERISTICS:
Population: Any intervention was indeed an arm that included each sub arm of different types of message that we tested against a control and pre-specified in our study protocol and analysis plan to combine arms for analysis.
Groups:
- Study Participants - Control: Study participants who are assigned to a pure control group
- Study Participants - Any Intervention: Study participants who are assigned to any intervention groups
- Total: Total of all reporting groups
Arm/Group | Study Participants - Control | Study Participants - Any Intervention | Total
Number analyzed (Participants) | 1617 | 12527 | 14144
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.16 (15.6) | 38.9 (15.2) | 38.93 (15.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 943 | 7169 | 8112
  Male | 674 | 5358 | 6032
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American | 1042 | 7725 | 8767
  Latinx | 575 | 4802 | 5377
Region of Enrollment [Number; unit: participants]
  United States | 1617 | 12527 | 14144
Household size [Mean (Standard Deviation); unit: person] | 3.23 (1.7) | 3.21 (1.7) | 3.22 (1.7)
Education index [Mean (Standard Deviation); unit: scores on a scale] — Education index is an integer capturing the highest level of education attained scored on a scale of 1 (third grade or less) to 11 (doctorate).
  scores on a scale | 4.53 (1.5) | 4.57 (1.5) | 4.56 (1.5)
Likely to run out of money because of COVID-19 [Count of Participants; unit: Participants] | 875 | 6531 | 7406
Trouble paying for food [Count of Participants; unit: Participants] | 558 | 4592 | 5150
Stratum [Count of Participants; unit: Participants]
  Female, age ≥45 y, coastal | 164 | 1154 | 1318
  Female, age ≥45 y, central | 229 | 1784 | 2013
  Female, age ≤44 y, coastal | 223 | 1787 | 2010
  Female, age ≤44 y, central | 327 | 2444 | 2771
  Male, age ≥45 y, coastal | 96 | 724 | 820
  Male, age ≥45 y, central | 111 | 885 | 996
  Male, age ≤44 y, coastal | 199 | 1740 | 1939
  Male, age ≤44 y, central | 268 | 2009 | 2277
Hispanic origin [Count of Participants; unit: Participants] — Population: The "Hispanic Origin" question is only applicable to Latinx participants.
  Participants
    number analyzed (Participants) | 575 | 4802 | 5377
    Mexican, Mexican American, Chicano | 387 | 3271 | 3658
    Cuba | 22 | 208 | 230
    Argentina | 8 | 74 | 82
    Colombia | 8 | 97 | 105
    Ecuador | 9 | 38 | 47
    El Salvador | 8 | 76 | 84
    Guatemala | 3 | 40 | 43
    Nicaragua | 5 | 19 | 24
    Panama | 2 | 20 | 22
    Peru | 8 | 55 | 63
    Spain | 27 | 189 | 216
    Venezuela | 9 | 50 | 59
    Other country | 73 | 608 | 681
    Puerto Rico | 6 | 57 | 63

OUTCOME MEASURES:

1. Primary Outcome: Incidence Rate for Knowledge Gaps: Control vs. Any Intervention
Description: Incidence rate for knowledge gaps is the count of knowledge gaps divided by the maximum possible count: 7
Time Frame: The outcome was measured immediately following the intervention in the 15-minute baseline survey.
Population: as for baseline characteristics
Measure: Mean (95% Confidence Interval); unit: proportion of knowledge gaps
Arm/Group | Study Participants - Control | Study Participants - Any Intervention
Number analyzed (Participants) | 1525 | 10711
proportion of knowledge gaps | 0.085 [0.076 to 0.093] | 0.065 [0.062 to 0.068]

2. Primary Outcome: Incidence Rate for Information-seeking Behavior: Control vs. Any Intervention
Description: Incidence rate for Information-seeking behavior is the count of links demanded divided by the maximum possible count: 10
Time Frame: The outcome was measured immediately following the intervention in the 15-minute baseline survey.
Population: as for baseline characteristics
Measure: Mean (95% Confidence Interval); unit: proportion of links
Arm/Group | Study Participants - Control | Study Participants - Any Intervention
Number analyzed (Participants) | 1450 | 10244
proportion of links | 0.335 [0.318 to 0.352] | 0.344 [0.338 to 0.351]

3. Primary Outcome: Incidence Rate for Knowledge Gaps by Intervention
Description: Incidence rate for knowledge gaps is the count of knowledge gaps divided by the maximum possible count: 7
Time Frame: The outcome was measured immediately following the intervention in the 15-minute baseline survey.
Population: Each intervention indicated in Arm/Group Title was indeed an arm that included each sub arm of different types of message that we tested Arm A against Arm B, or vice versa, and pre-specified in our study protocol and analysis plan to combine arms for analysis. Arms A and B are indicated in each Arm/Group Title.
Measure: Mean (95% Confidence Interval); unit: proportion of knowledge gaps
Groups:
- Intervention 1: Racial Discordance/Concordance Between Physician and Participant-Discordant (Arm A): Study participants who were assigned to receive an intervention of racial discordance between physician and participant.
- Intervention 1: Racial Discordance/Concordance Between Physician and Participant-Concordant (Arm B): Study participants who were assigned to receive an intervention of racial concordance between physician and participant.
- Intervention 2: Video 2 Recorded by MGH Physician/Dr. Birx of the CDC - MGH Physician (Arm A): Participants who were assigned to receive the social distancing component of the message is recorded by the MGH physicians.
- Intervention 2: Video 2 Recorded by MGH Physician/Dr. Birx of the CDC - Dr. Birx of the CDC (Arm B): Participants who were assigned to receive the social distancing component of the message is delivered by Dr. Birx of the CDC.
- Intervention 3: Received Acknowledgment of Discrimination - No (Arm A): Participants who were NOT assigned to receive the message include an acknowledgment of "elephant in the room" issues for each target group: trust in the medical system (African American participants) or fear of deportation (for Latinx participants)
- Intervention 3: Received Acknowledgment of Discrimination - Yes (Arm B): Participants who were assigned to receive the message include an acknowledgment of "elephant in the room" issues for each target group: trust in the medical system (African American participants) or fear of deportation (for Latinx participants)
- Intervention 4: Received Acknowledgment of Economic Inequalities - No (Arm A): Participants who were NOT assigned to receive the message acknowledged economic hardships that were associated with tight living quarters and working in essential services.
- Intervention 4: Received Acknowledgment of Economic Inequalities - Yes (Arm B): Participants who were assigned to receive the message acknowledged economic hardships that were associated with tight living quarters and working in essential services.
- Intervention 5: Received Information About Social Perception - No (Arm A); Intervention 5: Received Information About Social Perception - Yes (Arm B): Participants who were assigned to receive information about how representative individuals perceive mask wearers of color.
Arm/Group | Intervention 1: Racial Discordance/Concordance Between Physician and Participant-Discordant (Arm A) | Intervention 1: Racial Discordance/Concordance Between Physician and Participant-Concordant (Arm B) | Intervention 2: Video 2 Recorded by MGH Physician/Dr. Birx of the CDC - MGH Physician (Arm A) | Intervention 2: Video 2 Recorded by MGH Physician/Dr. Birx of the CDC - Dr. Birx of the CDC (Arm B) | Intervention 3: Received Acknowledgment of Discrimination - No (Arm A) | Intervention 3: Received Acknowledgment of Discrimination - Yes (Arm B) | Intervention 4: Received Acknowledgment of Economic Inequalities - No (Arm A) | Intervention 4: Received Acknowledgment of Economic Inequalities - Yes (Arm B) | Intervention 5: Received Information About Social Perception - No (Arm A) | Intervention 5: Received Information About Social Perception - Yes (Arm B)
Number analyzed (Participants) | 5395 | 5316 | 8041 | 2670 | 8010 | 2701 | 8058 | 2653 | 5366 | 5345
proportion of knowledge gaps | 0.066 [0.061 to 0.070] | 0.065 [0.061 to 0.069] | 0.065 [0.061 to 0.068] | 0.068 [0.061 to 0.074] | 0.066 [0.063 to 0.070] | 0.063 [0.057 to 0.069] | 0.066 [0.063 to 0.070] | 0.063 [0.057 to 0.069] | 0.066 [0.062 to 0.071] | 0.065 [0.060 to 0.069]

4. Primary Outcome: Incidence Rate for Information-seeking Behavior by Intervention
Description: as for outcome 2
Time Frame: The outcome was measured immediately following the intervention in the 15-minute baseline survey.
Population: as for outcome 3
Measure: Mean (95% Confidence Interval); unit: proportion of links
Arm/Group | Intervention 1: Racial Discordance/Concordance Between Physician and Participant-Discordant (Arm A) | Intervention 1: Racial Discordance/Concordance Between Physician and Participant-Concordant (Arm B) | Intervention 2: Video 2 Recorded by MGH Physician/Dr. Birx of the CDC - MGH Physician (Arm A) | Intervention 2: Video 2 Recorded by MGH Physician/Dr. Birx of the CDC - Dr. Birx of the CDC (Arm B) | Intervention 3: Received Acknowledgment of Discrimination - No (Arm A) | Intervention 3: Received Acknowledgment of Discrimination - Yes (Arm B) | Intervention 4: Received Acknowledgment of Economic Inequalities - No (Arm A) | Intervention 4: Received Acknowledgment of Economic Inequalities - Yes (Arm B) | Intervention 5: Received Information About Social Perception - No (Arm A) | Intervention 5: Received Information About Social Perception - Yes (Arm B)
Number analyzed (Participants) | 5147 | 5097 | 7697 | 2547 | 7653 | 2591 | 7696 | 2548 | 5142 | 5102
proportion of links | 0.336 [0.327 to 0.346] | 0.353 [0.343 to 0.362] | 0.343 [0.336 to 0.351] | 0.348 [0.335 to 0.362] | 0.346 [0.338 to 0.353] | 0.341 [0.328 to 0.354] | 0.344 [0.337 to 0.352] | 0.345 [0.332 to 0.358] | 0.345 [0.336 to 0.355] | 0.344 [0.334 to 0.353]

ADVERSE EVENTS:
Time Frame: 14 days
Arm/Group | Control - CDC - Mask (Control) - Concordant | Control - CDC - Mask (Control) - Discordant | Control - MGH - Mask (Control) - Concordant | Control - MGH - Mask (Control) - Discordant | Ack. Discrimination- MGH - Mask (Control) - Concordant | Ack. Discrimination- MGH - Mask (Control) - Discordant | Ack. Econ. Circumstance- MGH - Mask (Control ) Concordant | Ack. Econ. Circumstance - MGH - Mask (Control ) Discordant | Control Intro - CDC - Mask (antiStigma) Concordant | Control Intro - CDC - Mask (antiStigma) Discordant | Control - MGH - MaskS (antiStigma) Concordant Messenger | Control- MGH-MaskS (antiStigma) Discordant Messenger | Ack. Discrimination - MGH - MaskS (antiStigma) Concordant | Ack. Discrimination - MGH - MaskS (antiStigma) Discordant | Ack. Econ Hardship- MGH - Mask (antiStigma) Concordant | Ack. Econ Hardship- MGH - Mask (antiStigma) Discordant | Info Later - Pure Control
All-Cause Mortality (participants affected / at risk) | 0/784 | 0/791 | 0/780 | 0/778 | 0/777 | 0/788 | 0/783 | 0/788 | 0/779 | 0/780 | 0/782 | 0/790 | 0/779 | 0/786 | 0/781 | 0/781 | 0/1617
Serious Adverse Events (participants affected / at risk) | 0/784 | 0/791 | 0/780 | 0/778 | 0/777 | 0/788 | 0/783 | 0/788 | 0/779 | 0/780 | 0/782 | 0/790 | 0/779 | 0/786 | 0/781 | 0/781 | 0/1617
Other Adverse Events (participants affected / at risk) | 0/784 | 0/791 | 0/780 | 0/778 | 0/777 | 0/788 | 0/783 | 0/788 | 0/779 | 0/780 | 0/782 | 0/790 | 0/779 | 0/786 | 0/781 | 0/781 | 0/1617

LIMITATIONS AND CAVEATS:
Participants' behavior was not directly observed, outcomes were measured immediately postintervention in May 2020, and online recruitment may not be representative.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-14): https://cdn.clinicaltrials.gov/large-docs/19/NCT04371419/Prot_SAP_001.pdf